CLINICAL TRIAL: NCT05270512
Title: Evaluation of the Dermal Cooling System for Treatment of Common Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-21-001
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with Dermal Cooling System (Experimental): Dermal Cooling System will be used in all eligible subjects.
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Controlled localized cooling may be applied to lesions using the Dermal Cooling System.

SUMMARY:
The purpose of this study is to evaluate whether the Dermal Cooling System can be used to elicit an improvement in the cosmetic appearance or physical symptoms of common skin conditions.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label study to evaluate the effectiveness of the Dermal Cooling system to determine if cosmetic benefits or physical symptoms are achieved in common skin conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has a skin condition amenable to cryosurgical treatment including, for example, psoriasis, atopic dermatitis, acne, rosacea, and melasma.
3. Subject is willing to have skin exposed to cooling with the Dermal Cooling System.
4. Subject is willing to have digital photographs taken of the treatment area and agrees to use of photographs for presentation, educational, or marketing purposes.
5. Subject is willing to cover treated area or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area for the duration of the study, including the follow-up period, if requested.
6. Subject has read and signed a written informed consent form.
7. Subject is willing to comply with adjuvant topical regimen, as applicable.
8. Subject agrees not to undergo any other procedure(s) in the treatment area during the study.

Exclusion Criteria:

1. Dermatological conditions (e.g. vitiligo, open wounds, infection, pre-cancerous or malignant lesions) in the location of the treatment sites that would, in the professional opinion of the investigator, potentially pose an increased risk to the subject
2. Use of Accutane within the previous 6 months
3. History of melanoma
4. Subject is pregnant or intending to become pregnant during the study period
5. Subject is lactating or has been lactating in the past 6 months
6. Known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease.
7. History of abnormal wound healing or abnormal scarring
8. Inability or unwillingness to comply with the study requirements.
9. Current enrollment in a clinical study of any other unapproved investigational drug or device.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change in appearance in the treated area as determined by the Physician Global Assessment (PGA). | up to 3 months
  Investigator assessment using Physician Global Assessment (PGA); graded from "4" (very much improved") to "0" (worse).
Incidence of treatment-emergent adverse events | Up to 12 months
  The safety of the treatment is determined by the incidence of device- or procedure-related serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Tatsutani, PhD, Study Director — R2 Technologies
Locations (4):
- United States (4):
  - West Coast Research, Dublin, California
  - Oak Dermatology, Naperville, Illinois
  - Skin Search of Rochester, Inc., Rochester, New York
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No